CLINICAL TRIAL: NCT06348498
Title: A Open Label, Standardise-loaded and Single-Centre Phase Ⅰb Clinical Trial：Pharmacokinetic and Pharmacodynamic of Jia Shen Tablets in Chronic Heart Failure
Brief Title: Pharmacokinetic and Pharmacodynamic of Jia Shen Tablets in Chronic Heart Failure
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Tasly Pharmaceutical Group Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TSL-TCM-JSP-Ⅰb
Record Dates: First submitted 2024-03-12; First posted 2024-04-04 (Actual); Last update posted 2024-06-28 (Actual); Status verified 2024-03

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment Group (Experimental): Jia Shen Tablet，4 tablets，take orally，2 times a day
  Interventions: Drug: Jia Shen Tablet

INTERVENTIONS:
Drug: Jia Shen Tablet — Jia Shen Tablets contain 4 tablets (0.47 g per tablet), take orally, 2 times a day for 12 weeks

SUMMARY:
Evaluate the pharmacokinetic and pharmacodynamic characteristics of Jia Shen Tablets in patients with Chronic Heart Failure.

DETAILED DESCRIPTION:
Jia Shen Tablets are oral, compound traditional chinese medicine. This open label, standardise-loaded and single-Centre phase Ⅰb clinical trial will evaluate the pharmacokinetic and pharmacodynamic characteristics of Jia Shen Tablets in treatment of coronary heart disease complicating chronic heart failure (syndrome of Yang deficiency with blood stasis) and preliminarily evaluate the efficacy and safety.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75 years, either sex;
* Meet the diagnostic criteria for CHD and CHF;
* Meet the TCM differentiation criteria of yang deficiency and blood stasis in CHF;
* LVEF < 40% (Modified Simpson's Method);
* Class II to IⅢ for NYHA functional classification;
* Receive Steady dose of standard medication for CHF for at least 2 weeks;
* Understand the research requirements and are willing to provide written informed consent.

Exclusion Criteria:

* Acute heart failure or acute exacerbation of chronic heart failure;
* HF caused by other heart diseases, such as congenital heart disease, severe stenosis or insufficiency of heart valves, cardiomyopathy (e.g., hypertrophic obstructive cardiomyopathy, restrictive cardiomyopathy, dilated cardiomyopathy, alcoholic cardiomyopathy), moderate massive pericardial effusion, constrictive pericarditis, infective endocarditis;
* Patients with acute coronary syndrome within 30 days before receiving the trial drug，and the following situation within 6 months before receiving the trial drug，such as acute myocardial infarction，revascularization (e.g., PCI, CABG) or left ventricular reconstruction surgery, pacemaker implantation for cardiac resynchronization, and undergoing cardiothoracic surgery;
* Expect to receive an implantable device (e.g. ICD, CRT), or revascularization (e.g. PCI, CABG), or other cardiovascular surgery during the trial period;
* Severe arrhythmias [e.g., ventricular tachycardia, second degree type II or higher sinus or atrioventricular block without pacemaker placement, QT interval (QTc) greater than 480 ms after heart rate adjustment according to Fridericia's formula, or known history or symptoms of long QT syndrome];
* Combined with serious diseases of other systems, such as liver, kidney, hematopoietic system and other serious primary diseases, tumors, mental diseases, etc;
* The presence of uncontrolled hypertension (systolic blood pressure ≥180 mmHg and/or diastolic blood pressure ≥110 mmHg), or the presence of hypotension (systolic blood pressure < 80 mmHg and/or diastolic blood pressure < 50 mmHg);
* ALT or AST more than 3 times the upper limit of normal, and/or estimated glomerular filtration rate (eGFR) < 30 ml/min/1.73m2;
* Glycosylated hemoglobin (HbA1c) ≥9.0%, or fasting blood glucose ≥13.9 mmol/L;
* Anemia (Hb < 110 g/L for women, Hb < 120 g/L for men);
* Blood potassium is above the upper limit of normal;
* Patients who tested positive for five hepatitis B tests (except surface antibodies) or hepatitis C, or anti-TP or HIV antibodies;
* Patients with a history of drug abuse who test positive for drug abuse (morphine, methamphetamine, ketamine, dimethyldioxyamphetamine, THC, cocaine);
* Women who are pregnant or nursing, or have a need to have children within 3 months after the last dose of the trial;
* Participating in other studies and taking investigational drugs from other studies within 3 months prior to screening;
* Allergic to Jiashen tablets or their ingredients;
* Other situations judged by the researchers to be inappropriate for this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2024-04-09 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetic characteristic evaluation：Maximum observed plasma concentration (Cmax) | Day 1,27-30,56,84.
  To characterize the multiple dose PK of Jia Shen Tablets and assess the time required to reach steady state, the degree of accumulation and the time dependency of the PK in patients with Coronary Heart Disease Complicating Chronic Heart Failure (Syndrome of Yang Deficiency with Blood Stasis).
Plasma PK analysis: Time to reach peak or maximum observed concentration following drug administration (Tmax) | Day 1,27-30,56,84.
  To characterize the multiple dose PK of Jia Shen Tablets and assess the time required to reach steady state, the degree of accumulation and the time dependency of the PK in patients with Coronary Heart Disease Complicating Chronic Heart Failure (Syndrome of Yang Deficiency with Blood Stasis).
Plasma PK analysis: Area under curve at steady state (AUCss) | Day 1,27-30,56,84.
  To characterize the multiple dose PK of Jia Shen Tablets and assess the time required to reach steady state, the degree of accumulation and the time dependency of the PK in patients with Coronary Heart Disease Complicating Chronic Heart Failure (Syndrome of Yang Deficiency with Blood Stasis).

SECONDARY OUTCOMES:
NT-proBNP | Baseline to weeks 4,8 and 12.
  Change from baseline to weeks 4,8 and 12 in NT-proBNP.
6-Minutes-Walking-Test (6MWT) | Baseline to weeks 4,8 and 12.
  Change from baseline to weeks 4,8 and 12 in exercise capacity as measured by the 6-Minutes-Walking-Test (6MWT) distance.
Echocardiogram results | Baseline to weeks 12.
  Change from baseline to weeks 12 in left ventricular end diastolic diameter(LVEDD) measured by echocardiography.
  Change from baseline to weeks 12 in left ventricular end diastolic volume(LVEDV) measured by echocardiography.
  Change from baseline to weeks 12 in left ventricular end systolic volume(LVESV) measured by echocardiography.
  Change from baseline to weeks 12 in left ventricular ejection fraction(LVEF) measured by echocardiography.
  Change from baseline to weeks 12 in stroke volume(SV) measured by echocardiography.
  Change from baseline to weeks 12 in cardiac output(CO) measured by echocardiography.
NYHA classification | Baseline to weeks 4,8 and 12.
  Percentage of subjects whose NYHA classification improved/worsened/remained unchanged from baseline to weeks 4,8 and 12.
AEs | From baseline (Day1) till follow-up visit (Up to 12 week).
  Number of participants with adverse events (AEs).

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital of Tianjin University of Traditional Chinese Medicine, Tianjin, Tianjin Municipality, China